CLINICAL TRIAL: NCT04079816
Title: Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00025
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-20087
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- INVSENSOR00025 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00025 sensor.
  Interventions: Device: INVSENSOR00025

INTERVENTIONS:
Device: INVSENSOR00025 — Noninvasive pulse oximeter sensor

SUMMARY:
ORi is a unitless index that could help clinicians with their assessments or normoxic and hyperoxic states by scaling the measured absorption information between 0.00 and 1.00. An ORi of 0.00 corresponds to PaO2 values of 100mmHg and below and an ORi of 1.00 corresponds to PaO2 values of 200mmHg and above. In this study, the PaO2 is varied by controlling the concentration of oxygen the study volunteer breathes. Changes in ORi values are analyzed by comparing it to corresponding changes in PaO2 measurements from blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-50 years of age.
* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Carbon monoxide (CO) value less than or equal to 2.0% fractional carboxyhemoglobin (FCOHb).
* Subject has a physical status of ASA I or II (American Society of Anesthesiology Class 1; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Blood Pressure: (Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥50 mmHg), and if blood pressure is lower than 100/60 subject passes an orthostatic blood pressure test
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria: (*= Per physician discretion)

* Subject is pregnant.
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject smokes one pack of cigarettes or more in one week, and/or the equivalent of e-cigarette liquid, and smokers are not being recruited as indicated in the CSRF.
* Subject has open wounds, inflamed tattoos or piercings and/or any visible healing wounds that a medical professional renders them at an increased risk for participation.*
* Subject has known drug or alcohol abuse or uses recreational drugs.
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject who has taken anticoagulant medications within the last 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS).
* Subject has donated blood within the past 4 weeks.
* Subject has any chronic bleeding disorder (i.e. hemophilia)
* Subject has any symptomatic cardiac dysrhythmia (i.e. atrial fibrillation) and has not received clearance from their physician to participate.
* Subject has Wolff-Parkinson-White Syndrome or Stokes - Adams syndrome.
* Subject has known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's disease) that interferes with the subjects' level of consciousness.
* Subject has taken opioid pain medication within 24 hours of start of study.
* Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.).
* Subject is taking medications known to treat any type of infectious disease.*
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery*, appendix*, plastic surgery*.
* Subject has had invasive surgery within the past year- including but not limited to gallbladder, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has symptoms of congestion, head cold, flu or other illnesses.
* Subject is claustrophobic and/or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
* Subject has any cancer or history of cancer (not including skin cancer).*
* Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent Diabetes, or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the past 6 months.
* Subject intends to participate in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involved an arterial line.
* Subject has any medical condition which in the judgement of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator/study staff).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of of the 54 enrolled participants, 29 met inclusion criteria and proceeded to the study. The remainder of the enrolled participants include screen failures and subjects that did not proceed due to time constraints.
Period: Overall Study
Arm/Group | INVSENSOR00025
Started | 29
Completed | 26
Not Completed | 3
Not completed — Request of Subject | 2
Not completed — Unable to draw samples | 1

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00025
Number analyzed (Participants) | 26
Age, Customized [Count of Participants; unit: Participants]
  <18 years old | 0
  18 to 50 years old | 26
  >50 years old | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
  Hispanic | 8
  Asian or Pacific Islander | 4
  Black/Dark Skinned/African American | 7
  Middle Eastern | 1

OUTCOME MEASURES:

1. Primary Outcome: Concordance for Changes in ORi Values as Compared to Corresponding Changes in PaO2 Values.
Description: ORi is an index value without a unit and ORi does not directly measure PaO2. Therefore, sensitivity, specificity, and concordance are calculated to evaluate changes in ORi relative to the changes in PaO2.
Time Frame: 1-5 hours per subject
Measure: Number; unit: percentage of accuracy
Arm/Group | INVSENSOR00025
Number analyzed (Participants) | 26
percentage of accuracy
  PaO2 Threshold: 110 mmHg | 99.68
  PaO2 Threshold: 150 mmHg | 92.94
  PaO2 Threshold: 190 mmHg | 91.48

2. Primary Outcome: Specificity for Changes in ORi Values as Compared to Corresponding Changes in PaO2 Values.
Description: as for outcome 1
Time Frame: 1-5 Hours per subject
Measure: Number; unit: percentage of true negatives
Arm/Group | INVSENSOR00025
Number analyzed (Participants) | 26
percentage of true negatives
  PaO2 Threshold: 110 mmHg | 99.68
  PaO2 Threshold: 150 mmHg | 91.89
  PaO2 Threshold: 190 mmHg | NA — Changes in ORi (DeltaORi) are being compared to changes in PaO2 (DeltaPaO2 )in the reference PaO2 range of 100-200 mmHg. For the PaO2 threshold of 190 mmHg, reference PaO2 samples are outside the level of detection and thus data is not available to compute specificity.

3. Primary Outcome: Sensitivity for Changes in ORi Values as Compared to Corresponding Changes in PaO2 Values.
Description: as for outcome 1
Time Frame: 1 to 5 hours per subject
Measure: Number; unit: percentage of true positives
Arm/Group | INVSENSOR00025
Number analyzed (Participants) | 26
percentage of true positives
  PaO2 Threshold: 110 mmHg | NA — Changes in ORi (DeltaORi) are being compared to changes in PaO2 (DeltaPaO2 )in the reference PaO2 range of 100-200 mmHg. For the PaO2 threshold of 110 mmHg, reference PaO2 samples are outside the level of detection and thus data is not available to compute sensitivity.
  PaO2 Threshold: 150 mmHg | 93.67
  PaO2 Threshold: 190 mmHg | 91.78

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | INVSENSOR00025
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT04079816/Prot_SAP_000.pdf